CLINICAL TRIAL: NCT01277770
Title: Studies of Kidney Transplant Outcome
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 00011652
Record Dates: First submitted 2010-08-19; First posted 2011-01-17 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Transplant Recipient (Kidney); Steroid-Free Maintenance Immunosuppression; Post-Transplant Infections; Thymoglobulin
Keywords: Thymoglobulin; Kidney Transplant Recipients; Steroid-Free; Immunosuppression
MeSH Terms: interventions — Immunosuppression Therapy; Transplantation; thymoglobulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney Transplant Recipients: Kidney Transplant Recipients at the University of Minnesota since 1984. The study looks at a 10 year followup of steroid-free maintenance immunosuppression, post-transplant infections and evaluation of the DGF nomogram in Thymoglobulin on patients at the University of Minnesota.
  Interventions: Drug: Steroid-Free Maintenance Immunosuppression; Other: Infection After Kidney Transplantation; Drug: Evaluation of the DGF nomogram in Thymoglobulin

INTERVENTIONS:
Drug: Steroid-Free Maintenance Immunosuppression — 10 year follow-up of steroid-free maintenance immunosuppression
  Other Names: Steroid-Free; Immunosuppression
Other: Infection After Kidney Transplantation — A cross-sectional study of infection after kidney transplantation (with emphasis on infection in steroid-free recipients).
  Other Names: Infection; Transplantation; Steroid-Free
Drug: Evaluation of the DGF nomogram in Thymoglobulin — An evaluation of the DGF nomogram in Thymoglobulin treated recipients at the University of Minnesota
  Other Names: Thymoglobulin

SUMMARY:
The purpose of this study is to improve outcome for kidney transplant recipients. There has not been commensurate improvement in medium and long-term outcomes. Ongoing clinical research is necessary to improve transplant outcomes.

DETAILED DESCRIPTION:
This study is looking at information already collected of transplant outcomes (short, medium and long-term complications and quality of life). This will specifically look at:

1. 10 year follow-up of steroid-free maintenance immunosuppression
2. A cross-sectional study of infection after kidney transplantation (with emphasis on infection in steroid-free recipients
3. An evaluation of the Delayed Graft Function (DGF) nomogram in Thymoglobulin treated recipients at the University of Minnesota

ELIGIBILITY:
Inclusion Criteria:

* Kidney Transplant Recipient at the University of Minnesota
* Kidney Transplant Recipients on steroid-free maintenance immunosuppression

Exclusion Criteria:

* Non-kidney transplant patients at the University of Minnesota

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients at the University of Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2009-05; Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Data Analysis | 10 year followup
  All studies are analyses from the Transplant Outcomes Database. Recipients have signed consent to have medical information entered into the database for these analyses. The database contains information on short, medium and long-term results.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Matas, MD, Principal Investigator — University of Minnesota
Locations (1):
- University Of Minnesota, Minneapolis, Minnesota, United States